CLINICAL TRIAL: NCT03328117
Title: A Randomized, Placebo-controlled, Double-blind Study to Investigate the Effects of the Tyrosine Kinase Inhibitor Imatinib on Pulmonary Vascular Dysfunction in a Human Experimental Model of Acute Lung Injury
Brief Title: A Study to Investigate the Effects of Imatinib on Pulmonary Vascular Dysfunction in a Human Model of Lung Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exvastat Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXV001; 2017-002203-10 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Drug: Imatinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Imatinib — Over-encapsulated 100 mg imatinib mesilate tablets
  Arms: Intervention
Drug: Placebo oral capsule — Matching placebo oral capsule
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled clinical study of imatinib (as mesilate) in healthy subjects exposed inhaled lipopolysaccharide. During the study, eight oral doses of imatinib, or placebo, will each be taken 12 hours apart, before subjects are exposed to nebulized lipopolysaccharide (LPS). Four hours after LPS exposure, a bronchoalveolar lavage (BAL) will be undertaken, and BAL fluid (BALF collected. Once study assessments are completed, a follow-up visit will be conducted approximately 7 days after the last dose of imatinib.

The primary objective of the study is to investigate the effect of imatinib on LPS-induced pulmonary vascular dysfunction. The primary endpoints of this study are:

1. Change in the number of neutrophils in BALF 6 hours after the LPS challenge in subjects exposed to imatinib compared with placebo.
2. Change in concentration of total protein in BALF 6 hours after the LPS challenge in subjects exposed to imatinib compared with placebo

ELIGIBILITY:
Inclusion Criteria:

1. Are able and willing to provide written informed consent to participate in this clinical study.
2. Healthy males and females, between 18 and 55 years old (both inclusive) at the screening visit.
3. Male subjects must practice an acceptable contraceptive method from the time of first IMP administration until 6 weeks after the follow-up visit.
4. Female subjects must either be:

   1. Of non-childbearing potential:
   2. Or if of childbearing potential, must practice an acceptable contraceptive method from 4 weeks before the first IMP administration until 6 weeks after the follow-up visit.
5. Good general health as ascertained by detailed medical history and physical examination at the screening visit.
6. Body mass index ≥18.0 and ≤30 kg/m2 at the screening visit.
7. No clinically relevant abnormalities in the 12-lead ECG as per the Investigator's judgement at the screening visit
8. No clinically relevant abnormalities in results of clinical laboratory tests as per the Investigator's judgement at the screening visit.
9. Normal spirometry (FEV1 ≥ 85% of predicted, FEV1/FVC ratio ≥ 70%) at the screening visit.
10. Non-smokers or no history of smoking (including e-cigarettes and other forms of vaporizing/inhalation) in the last 6 months prior to the screening visit.
11. Subjects must be able to communicate well with the Investigator/designee.

Exclusion Criteria:

1. History of hypersensitivity to the IMP or any of the excipients or to medicinal products with similar chemical structures.
2. Presence of any clinically relevant acute or chronic disease which could interfere with the subject safety during the study, expose the subject to undue risk, limit the biological sampling, interfere with the absorption of the investigational product (or interfere with the study objectives.
3. Any history of previous respiratory, hematological or malignant disease, including childhood asthma.
4. Any history of chronic renal, cardiac (previous myocardial infarction, diagnosis of cardiac failure or cardiac rhythm disturbances such as atrial fibrillation) or hepatic impairment.
5. Current evidence of ongoing or acute infection, history of repeated or chronic significant infections, or history of serious infection within 3 months of randomization. Acute infection is defined as a history of febrile illness (> 38°C), or 2 or more of the following symptoms within the last 7 days prior to the screening visit or Day 1: cough, sore throat, runny nose, sneezing, limb/joint pain, headache or vomiting/diarrhea.
6. Any condition that in the opinion of the Investigator will require regular concomitant medication including herbal products, or predicted need of any concomitant medication during the study.
7. Intake of any prescription and over-the-counter medication (except paracetamol, hormonal contraceptives and hormonal replacement therapy) including herbal and dietary supplements (including St John's Wort), vitamins and minerals, within 7 days or 5 half-lives (whichever is longer) prior to the first dose of IMP.
8. Systolic blood pressure < 90 mmHg or > 140 mmHg, or diastolic blood pressure < 50 mmHg or > 90 mmHg after 5 minutes in the supine position at the screening visit.
9. Positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV)-1 and/or -2 antibodies at the screening visit.
10. Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee) or intake of food or drinks containing xantine (e.g., caffeine) within 24 hours prior to the screening visit or Day 1.
11. Positive urine cotinine test at the screening visit or Day 1, or the inability to stop using nicotine-containing products during the clinical study.
12. History or presence of drug addiction (positive urine drug screen at the screening visit or Day 1).
13. History of regular alcohol consumption within 6 months of the screening visit defined as an average weekly intake of > 21 units (or an average daily intake of > 3 units) for males or an average weekly intake of > 14 units (or an average daily intake > 2 units) for females.
14. Positive urine alcohol test at the screening visit or Day 1, or the inability to refrain from the use of alcohol during the clinical study.
15. Intake of any food or any drinks containing grapefruit, Chinese grapefruit (pomelo), Seville orange (including marmalade) or quinine-containing products (e.g., tonic water, bitter lemon) from 7 days prior to Day 1.
16. Blood component or plasma donation within 3 months prior to the first dose of IMP.
17. Participation in another study with an experimental drug within 3 months before the first dose of IMP. Exclusion period starts from last IMP dosed in previous study to first dose of IMP.
18. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent, or limited the ability of the subject to comply with the protocol requirements.
19. Subject is mentally or legally incapacitated.
20. A pregnant woman or a nursing mother.
21. Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude and improbability of completing the clinical study.
22. Subjects who, in the opinion of the Investigator, are considered unsuitable for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Change in the number of neutrophils in bronchoalveolar lavage fluid in subjects exposed to imatinib compared with placebo | 6 hours after lipopolysaccharide inhalation
  Change in the number of neutrophils in bronchoalveolar lavage fluid in subjects exposed to imatinib compared with placebo
Change in concentration of total protein in bronchoalveolar lavage fluid in subjects exposed to imatinib compared with placebo | 6 hours after the LPS challenge
  Change in concentration of total protein in bronchoalveolar lavage fluid in subjects exposed to imatinib compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBBCh, Principal Investigator — Parexel
Locations (1):
- PAREXEL Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No